CLINICAL TRIAL: NCT05552846
Title: Consolidative Thoracic Radiotherapy for Extensive-stage Small-cell Lung Cancer Treated with Chemo-immunotherapy Followed by PD-1/PD-L1 Maintenance Therapy：an Open Label, Single Arm Prospective Trial
Brief Title: Phase II Trial of Consolidative Thoracic Radiotherapy for ES-SCLC After Standard Care of Chemo-immunotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, QIWEIXIANG, Prof., Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021（212）
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-11

CONDITIONS: Small-cell Lung Cancer
Keywords: thoradic radiotherapy; immune checkpoint inhibitors; chemo-immunotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental group (Experimental): chemo-immunotherapy followed by thoracic radiotherapy and PD-1/PD-L1 maintenance therapy
  Interventions: Radiation: thoracic radiotherapy

INTERVENTIONS:
Radiation: thoracic radiotherapy — Four courses of carboplatin/etoposide/anti-PD-1/PD-L1 every 3 weeks All the enrolled patients will be patients with ES-SCLC who did not have PD (determined as per the RECIST v1.1) after 6 cycle of platinum-based chemotherapy in combination with an anti-PD-1/L1. Then, thoracic radiotherapy of 45 Gy/15 fractions. PD-1/PD-L1 maintenance therapy concurrently and after thoracic radiotherapy at least more than 6 months, or until intolerable toxicity, progressive disease leading to a need for other treatment, or until the patient no longer wishes to continue treatment.

SUMMARY:
This is an open-label, single arm Phase II study designed to evaluate the efficacy and safety of thoracic radiotherapy for extensive-stage small-cell lung cancer treated with PD-1/PD-L1 plus etoposide platinum followed by PD-1/PD-L1 maintenance therapy

DETAILED DESCRIPTION:
This study a single arm prospective phase II study. All the enrolled patients will be patients with ES-SCLC who did not have PD (determined as per the RECIST v1.1) after 6 cycle of platinum-based chemotherapy in combination with an anti-PD-1/L1. Then, those enrolled patients would be treated with thoracic radiotherapy concurrently with PD-1/PD-L1 maintenance therapy, and the total maintenance therapy time should at least more than 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age between18 years and 80 years at time of study entry
2. ECOG performance status of 0 or 1
3. Body weight >30 kg
4. Adequate bone marrow, liver and kidney function
5. Life expectancy of at least 3 months
6. At least one measurable (RECIST 1.1), thoracic lesion that can be irradiated with 45 Gy/15 fractions
7. Histologic or cytologic confirmation of small cell lung cancer
8. Stage III-IV disease (TNM v8)
9. Adequate pulmonary function with FEV1 >1 L or >30 % of predicted value and DLCO >30 % of predicted value
10. Patients with brain metastases are eligible provided they are asymptomatic or treated and stable on steroids and/or anticonvulsants prior to the start of treatment -

Exclusion Criteria:

1. Previous chemo-, immuno- or radiotherapy for SCLC
2. Major surgical procedure last 28 days
3. History of allogenic organ transplantation, autoimmune disease, immunodeficiency, hepatitis or HIV
4. Uncontrolled intercurrent illness
5. Other active malignancy
6. Leptomeningeal carcinomatosis
7. Immunosuppressive medication
8. Pregnant or breastfeeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2021-01-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
1-year progression-free survival | 12 months after last patient entry
  PFS is defined as the period from the start of receiving the first EC/EP chemotherapy plus PD-1/PD-L1 inhibitor to disease progression.

SECONDARY OUTCOMES:
1-year overall survival | 12 months after last patient entry
toxicities | 12 months after last patient entry
  Number of participants with treatment-related adverse events and the grade of adverse events as assessed by CTCAE v4.0
5-year overall survival | 5-year after last patient entry

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai jiaotong univestigy school of medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No